CLINICAL TRIAL: NCT06070623
Title: Role of Sonograpic Evaluation Via Doppler and Elastography in Evaluation of Hepatic Neoplasms Post TACE With Correlation With Modified RECIST Criteria.
Brief Title: Follow up After TACE by Elastography and Color Doppler.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marco Moheb Samaan Drota, Dr at diagnostic and interventional radiology department - South Egypt cancer institute, Assiut University
Other Study IDs: Elastography, Doppler in TACE.
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: US — We use elastography and color Doppler from US machine and compare results with CT
  Other Names: CT

SUMMARY:
To determine accuracy of elastography and color Doppler in follow up of patients with HCC after TACE comparing with modified RECIST criteria.

DETAILED DESCRIPTION:
The incidence of liver cancer is one of the highest in the world. In Egypt HCC is the forth common cancer and represents up to 90% of all liver malignancies. Where it is responsible for 33.63% and 13.54% of all cancers in males and females respectively.

Transarterial chemoembolization (TACE) is recommended as the first-line treatment in early stage patients with hepatocellular carcinoma (HCC) or as a palliative treatment modality in advanced patients with unresctable tumor which was known to increase survival rate. However, tumor control usually requires multiple TACE interventions due to the presence of residual and recurrent lesions.

Currently the Response Evaluation Criteria in Solid Tumors (RECIST) guideline was proposed as a method for measuring treatment response based on tumor shrinkage, which is a valuable measure of antitumor activity of cytotoxic drugs, Which adapted the concept of viable tumor-tumoral tissue showing uptake in arterial phase of contrast-enhanced MSCT abdomen.

Elastography can provide information about tumor stiffness to predict tumor response after TACE and detect any residual or recurrence.

We also use color Doppler in follow up to detect changes in portal pressure and hepatic artries hemodynamics of HCC patients after TACE. Mainly we search for changes in portal vein velocity {PVVel}, hepatic artery resistive index {HARI} and hepatic artery pulsitality index {HAPI}.

ELIGIBILITY:
Inclusion Criteria:

* All patients with hepatocellular carcinoma underwent TACE in South Egypt cancer institute.

Exclusion Criteria:

* Patients with liver metastases.
* Patients with hepatic or perihepatic inflammations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hepatic focal lesion , which is eligable to trans arterial chemoebmolization.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Role of elastography and color Doppler to follow up after TACE. | Baseline
  Accuracy of elastography and color Doppler in follow up of patients with HCC who underwent TACE, compared to modified RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Thabet, Prof Dr, Study Director — Professor doctor at radiology department - Assiut University; Haysam Samy, Prof Dr, Study Director — Professor doctor at radiology department - South Egypt cancer institute; Mohamed Elbaroudy, Ass. Prof Dr, Study Director — Assistant professor doctor at radiology department - South Egypt cancer institute

REFERENCES:
- [Background] Tierney J, Baker J, Borgmann A, Brown D, Byram B. Non-contrast power Doppler ultrasound imaging for early assessment of trans-arterial chemoembolization of liver tumors. Sci Rep. 2019 Sep 10;9(1):13020. doi: 10.1038/s41598-019-49448-8. PMID 31506503
- [Background] Sato Y, Watanabe H, Sone M, Onaya H, Sakamoto N, Osuga K, Takahashi M, Arai Y; Japan Interventional Radiology in Oncology Study Group-JIVROSG. Tumor response evaluation criteria for HCC (hepatocellular carcinoma) treated using TACE (transcatheter arterial chemoembolization): RECIST (response evaluation criteria in solid tumors) version 1.1 and mRECIST (modified RECIST): JIVROSG-0602. Ups J Med Sci. 2013 Mar;118(1):16-22. doi: 10.3109/03009734.2012.729104. Epub 2012 Nov 20. PMID 23167460
- [Background] Hou S, Hua S, Cui K, Liu F, Ding K, Yuan J. The course and prognostic value of tumor stiffness detected by ultrasound elastography for transarterial chemoembolization of hepatocellular carcinoma. Quant Imaging Med Surg. 2023 Jun 1;13(6):3962-3972. doi: 10.21037/qims-22-292. Epub 2023 May 9. PMID 37284088
- [Background] Conti CB, Cavalcoli F, Fraquelli M, Conte D, Massironi S. Ultrasound elastographic techniques in focal liver lesions. World J Gastroenterol. 2016 Mar 7;22(9):2647-56. doi: 10.3748/wjg.v22.i9.2647. PMID 26973405